CLINICAL TRIAL: NCT03773978
Title: A Randomized, Double-Blind, Placebo-Controlled, Withdrawal, Safety and Efficacy Study of Oral Baricitinib in Patients From 2 Years to Less Than 18 Years Old With Juvenile Idiopathic Arthritis (JIA)
Brief Title: A Study of Baricitinib in Participants From 2 Years to Less Than 18 Years Old With Juvenile Idiopathic Arthritis
Acronym: JUVE-BASIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16276; I4V-MC-JAHV (Other: Eli Lilly and Company); 2017-004518-24 (EudraCT Number)
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Polyarticular JIA; Oligoarthritis; Juvenile psoriatic arthritis (JPsA); Enthesitis-related juvenile idiopathic arthritis (ERA)
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Baricitinib was administered QD (once daily) as a 4-mg oral tablet for adolescent participants (12 to <18 years of age) and children ≥9 years of age; and 2 mg for children <9 years of age. Participants <6 years of age received an oral suspension. Participants ≥6 to <12 years old had the option of receiving an oral suspension. Participants >12 years old were supplied tablets. The oral suspension dose was administered as 4-mg, 2-mg, 1-mg, and 0.5-mg as needed.
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Placebo matched to baricitinib was administered to participants during the DBW period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally.
  Other Names: LY3009104
  Arms: Baricitinib
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the study drug baricitinib given orally is safe and effective in participants with JIA from 2 years to less than 18 years old.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have had a diagnosis of active JIA (polyarticular, extended oligoarticular, or enthesitis-related juvenile idiopathic arthritis [ERA] including JPsA).
* Participants must have had an inadequate response to at least one conventional or biologic disease-modifying antirheumatic drug (DMARD).

Exclusion Criteria:

* Participants must not have systemic JIA, with or without active systemic features.
* Participants must not have persistent oligoarticular arthritis.
* Participants must not have been previously treated with a Janus kinase (JAK) inhibitor.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (86):
- Argentina (3):
  - Instituto CAICI SRL, Rosario, Santa Fe Province
  - Centro Medico Privado de Reumatologia, SAN M. de Tucuman, Tucumán Province
  - Hospital General de Niños Dr. Pedro de Elizalde, Buenos Aires
- Australia (3):
  - The Sydney Children's Hospitals Network, Westmead, New South Wales
  - Royal Childrens Hospital Melbourne, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- Austria (2):
  - LKH Bregenz, Bregenz, Vorarlberg
  - AKH, Vienna
- Belgium (3):
  - UCL- Saint Luc, Brussels, Brussels Capital
  - UZ Gent-Reuma, Ghent, East Flanders
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Brazil (4):
  - CMIP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Faculdade de Ciências Médicas - UNICAMP, Campinas, São Paulo
  - Universidade Federal de São Paulo - Escola Paulista de Medicina, São Paulo
- China (5):
  - Children's hospital of Nanjing, Nanjing, Jiangsu
  - Children's Hospital of Chongqing Medical University, Chongqing, Tianjin City
  - Capitol Institute of Pediatrics Children'S Hospital, Beijing
  - Beijing Children's hospital, Capital Medical University, Beijing
  - Children's Hospital of Soochow University, Suzhou
- Czechia (2):
  - Centrum detske revmatologie VFN, Klinika detskeho a dorostoveho lekarstvi 1.LFUK a VFN v Praze, Prague
  - Fakultni Nemocnice v Motole, Prague
- Denmark (2):
  - Center for Børnereumatologi. Børn og Unge, Århus Universitetshospital, Århus N
  - Paediatric rheumatology Unit, København Ø
- France (5):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - GH Necker - Enfants Malades, Paris
  - CHU la Miletrie, Poitiers
- Germany (6):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Asklepios Klinik Sankt Augustin, Saint Augustin, North Rhine-Westphalia
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Charité Universitätsmedizin Berlin Campus Buch, Berlin
  - Schön Klinik Hamburg Eilbek, Hamburg
- India (3):
  - Sri Ramachandra MedicaL College & Research Institute, Porur, Chennai
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College Vellore, Vellore, Tamil Nadu
- Israel (4):
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Schneider Children's Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (7):
  - ASST Spedali Civili - Università degli Studi, Brescia
  - Ospedale SS. Annunziata, Chieti
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Ospedale Pediatrico Gaslini - Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Infantile Burlo Garofolo, Trieste
- Japan (11):
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Miyagi Children's Hospital, Sendai, Miyagi
  - Osaka Medical ＆ Pharma Univ Hp, Takatsuki, Osaka
  - Saitama Children's Medical Center, Saitama-shi, Saitama
  - Tokyo Medical And Dental University Medical Hospital, Bunkyō, Tokyo
  - St. Lukes International Hospital, Chuo-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Kagoshima University Hospital, Kagoshima
  - Niigata University Medical & Dental Hospital, Niigata
- Mexico (5):
  - Clinstile, S.A. de C.V., Cuauhtémoc, Federal District
  - CREA de Guadalajara, S.C., Guadalajara, Jalisco
  - Hospital Univ. "Dr. José Eleuterio González", Monterrey, Nuevo León
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C, Durango
- Poland (3):
  - Wojewódzki Specjalistyczny Szpital Dziecięcy im. św. Ludwika w Krakowie, Krakow
  - CSK, Uniwersyteckie Centrum Pediatrii im.M.Konopnickiej,Klinika Kardiologii i Reumatologii Dzieciecej, Lodz
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji, Warsaw
- Russia (5):
  - V.A. Nasonova Research Institute of Rheumatology, Moscow
  - Morozovsky Children's City Clinical Hospital, Moscow
  - First Moscow State Medical University n.a. Sechenov, Moscow
  - Scientific Center of Children's Health, Moscow
  - Saint-Petersburg State Pediatric Medical University, Saint Petersburg
- Spain (6):
  - Hospital Sant Joan de Deu, Barcelona, Catalonia
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Fe de Valencia, Valencia
- Turkey (Türkiye) (2):
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Dokuz Eylul University Hospital, Izmir
- United Kingdom (5):
  - University College Hospital - London, London, Greater London
  - Great Ormond Street Hospital For Children NHS Foundation Trust, Bloomsbury, London
  - Sheffield Children's Hospital, Sheffield, South Yorkshire
  - Bristol Royal Hospital for Children, Bristol
  - Alder Hey Children's NHS Foundation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Krishnan V, Keller SY, Chew C, Sims JT, Chang CY, Dow ER, Benschop RJ, Wang R, Ramanan AV. Serum biomarkers associated with baricitinib response in patients with juvenile idiopathic arthritis: a post-hoc analysis of the phase 3 JUVE-BASIS trial. Lancet Rheumatol. 2025 Nov;7(11):e799-e807. doi: 10.1016/S2665-9913(25)00153-5. Epub 2025 Sep 4. PMID 40915298
- [Derived] Ramanan AV, Quartier P, Okamoto N, Foeldvari I, Spindler A, Fingerhutova S, Anton J, Wang Z, Meszaros G, Araujo J, Liao R, Keller S, Brunner HI, Ruperto N; JUVE-BASIS investigators; Paediatric Rheumatology International Trials Organisation. Baricitinib in juvenile idiopathic arthritis: an international, phase 3, randomised, double-blind, placebo-controlled, withdrawal, efficacy, and safety trial. Lancet. 2023 Aug 12;402(10401):555-570. doi: 10.1016/S0140-6736(23)00921-2. Epub 2023 Jul 6. PMID 37423231
- See also: A Study of Baricitinib in Participants From 2 Years to Less Than 18 Years Old With Juvenile Idiopathic Arthritis — https://trials.lillytrialguide.com/en-US/trial/4q06tGZPTqsikCQMw0kcYI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 220 participants were enrolled: 29 started with the Pharmacokinetics (PK)/Safety period (2 weeks), and one participant was discontinued due to protocol deviation. 191 participants entered into the Open-label lead-in period (OLLI) period, and during week 2, 28 participants from the PK/Safety population entered into the OLLI period.
Pre-assignment Details: Participants entered the PK/Safety period (0 to 2 weeks) in staggered enrollment of 4 age groups (12 to <18, 9 to <12, 6 to <9, and 2 to <6 years). Upon the confirmation of the safety comparability assessment, remaining participants were enrolled directly into the OLLI period (0 to 12 weeks) followed by a double-blind randomised withdrawal placebo-controlled period (DBW) period (12 to 44 weeks) in which participants were randomized to baricitinib or placebo.
Groups:
- Baricitinib: Baricitinib was administered once daily (QD) as a 4-mg for adolescent participants (12 to <18 years of age) and children ≥9 years of age; and 2 mg for children <9 years of age. Participants <6 years of age received an oral suspension. Participants ≥6 to <12 years old had the option of receiving an oral suspension. Participants >12 years old were supplied tablets.
Period: PK/Safety and OLLI Period
Arm/Group | Baricitinib | Placebo
Started | 220 | 0
PK/Safety Period | 29 (One participant was discontinued from this period due to the protocol violation.) | 0
OLLI Period | 219 (191 participants entered into the Open-label lead-in period (OLLI) period, and during week 2, 28 participants from PK/Safety population entered into the OLLI period.) | 0
Received at Least One Dose of Study Drug | 220 | 0
Completed | 163 | 0
Not Completed | 57 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Failure to Meet Randomization Criteria | 39 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Due to epidemic or pandemic | 6 | 0
Not completed — unexplainable flare disease | 1 | 0
Not completed — Protocol Violation | 4 | 0
Not completed — Participant transitioned to JAHX | 1 | 0
Not completed — Investigational product was not delivered to the site | 1 | 0
Period: DBW Period
Arm/Group | Baricitinib | Placebo
Started | 82 (Participants who completed the OLLI period of the study were randomized to Baricitinib and placebo in DBW period.) | 81 (Participants who completed the OLLI period of the study were randomized to Baricitinib and placebo in DBW period.)
Completed | 56 | 32
Not Completed | 26 | 49
Not completed — Adverse Event | 2 | 2
Not completed — Failure to Meet Continuation Criteria | 16 | 40
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Due to epidemic or pandemic | 5 | 6
Not completed — Study team decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis Population includes all randomized participants.
Groups:
- Baricitinib: Baricitinib was administered QD (once daily) as a 4-mg for adolescent participants (12 to <18 years of age) and children ≥9 years of age; and 2 mg for children <9 years of age. Participants <6 years of age received an oral suspension. Participants ≥6 to <12 years old had the option of receiving an oral suspension. Participants >12 years old were supplied tablets.
Arm/Group | Baricitinib
Number analyzed (Participants) | 220
Age, Customized [Count of Participants; unit: Participants]
  Age: >=2 to <6 years | 6
  Age: >=6 to <9 years | 9
  Age: >=9 to <12 years | 30
  Age: >=12 to <18 years | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43
  Not Hispanic or Latino | 133
  Unknown or Not Reported | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 48
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 152
  More than one race | 2
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 20
  Czechia | 12
  Japan | 25
  United Kingdom | 11
  India | 6
  Spain | 14
  Russia | 8
  Austria | 2
  Turkey | 3
  Belgium | 7
  China | 18
  Brazil | 2
  Poland | 7
  Denmark | 1
  Italy | 11
  Mexico | 21
  Israel | 15
  France | 10
  Australia | 1
  Germany | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Flare
Description: A disease flare is defined as a worsening of 30% or more in at least three of the six core Paediatric American College of Rheumatology (PedACR) criteria for juvenile rheumatoid arthritis (JIA) and an improvement of 30% or more in no more than one of the criteria. The six PedACR criteria are: 1) the number of active joints, 2) the number of joints with limited range of motion, 3) physician's global assessment of disease activity, 4) parent's global assessment of the participant's overall well-being, 5) physical function as measured by the Childhood Health Assessment Questionnaire (CHAQ) and 6) acute-phase reactant (high-sensitivity C-reactive protein [hsCRP] and erythrocyte sedimentation rate [ESR]), the ESR measure is only used as an acute phase reactant in the core criteria.
Time Frame: Week 12 to Week 44
Population: DBW Population: All randomized participants from the DBW period who had data for time to disease flare at given time point.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Weeks | NA [NA to NA] — Median, upper and lower limits of 95% CI was not estimable due to small number of participants with the event. | 27.14 [15.29 to NA] — Upper limit of 95% CI was not estimable due to small number of participants with the event.
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.241, 95% CI 2-sided [0.128 to 0.453]

2. Secondary Outcome: Percentage of Participants Achieving PedACR30 Responder Index
Description: The PedACR30 response is defined as at least 30% improvement from baseline in 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by >30%. The 6 core response variables included in the PedACR criteria are: Number of active joints (defined as a joint that is swollen or in the absence of swelling has loss of passive motion accompanied by either pain on motion or joint tenderness) in 73 joints, Number of joints with limited range of motion in 69 joints, Physician's Global Assessment of Disease Activity (21-circle visual analogue scale [VAS]), Parent's Global Assessment of Patient's Overall Well-being, Physical function as assessed by the CHAQ and Acute-phase reactant (hsCRP and ESR). When PedACR response is analyzed as secondary endpoint, ESR measure is only used as acute-phase reactant in the core criteria.
Time Frame: Week 16, 20, 24, 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for PedACR30 at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 16 | 92.7 [87 to 98.3] | 81.5 [73 to 89.9]
  At week 20 | 87.8 [80.7 to 94.9] | 64.2 [53.8 to 74.6]
  At week 24 | 85.4 [77.7 to 93.0] | 55.6 [44.7 to 66.4]
  At week 28 | 78 [69.1 to 87] | 51.9 [41 to 62.7]
  At week 32 | 74.4 [64.9 to 83.8] | 49.4 [38.5 to 60.3]
  At week 36 | 72.0 [62.2 to 81.7] | 44.4 [33.6 to 55.3]
  At week 40 | 69.5 [59.5 to 79.5] | 38.3 [27.7 to 48.9]
  At week 44 | 67.1 [56.9 to 77.2] | 38.3 [27.7 to 48.9]
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; at week 16; Test type: Superiority; p = 0.052, Regression, Logistic; Odds Ratio (OR) = 2.72, 95% CI 2-sided [0.99 to 7.46]
Statistical Analysis 2: Comparison: Baricitinib vs Placebo; at week 20; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 3.64, 95% CI 2-sided [1.60 to 8.28]
Statistical Analysis 3: Comparison: Baricitinib vs Placebo; at week 24; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.34, 95% CI 2-sided [2.00 to 9.41]
Statistical Analysis 4: Comparison: Baricitinib vs Placebo; at week 28; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 3.37, 95% CI 2-sided [1.62 to 7.01]
Statistical Analysis 5: Comparison: Baricitinib vs Placebo; at week 32; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 3.00, 95% CI 2-sided [1.48 to 6.07]
Statistical Analysis 6: Comparison: Baricitinib vs Placebo; at week 36; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.25, 95% CI 2-sided [1.62 to 6.52]
Statistical Analysis 7: Comparison: Baricitinib vs Placebo; at week 40; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.70, 95% CI 2-sided [1.85 to 7.41]
Statistical Analysis 8: Comparison: Baricitinib vs Placebo; at week 44; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.27, 95% CI 2-sided [1.65 to 6.50]

3. Secondary Outcome: Percentage of Participants Achieving PedACR50 Responder Index
Description: The PedACR50 response is defined as at least 50% improvement from baseline in 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by > 30%. The 6 core response variables included in the PedACR criteria are: Number of active joints (defined as a joint that is swollen or in the absence of swelling has loss of passive motion accompanied by either pain on motion or joint tenderness) in 73 joints, Number of joints with limited range of motion in 69 joints, Physician's Global Assessment of Disease Activity (21-circle VAS), Parent's Global Assessment of Patient's Overall Well-being, Physical function as assessed by the CHAQ and Acute-phase reactant (hsCRP and ESR). When PedACR response is analyzed as secondary endpoint, ESR measure is only used as acute-phase reactant in the core criteria.
Time Frame: Week 16, 20, 24, 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for PedACR50 at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 16 | 79.3 [70.5 to 88] | 75.3 [65.9 to 84.7]
  At week 20 | 81.7 [73.3 to 90.1] | 58 [47.3 to 68.8]
  At week 24 | 81.7 [73.3 to 90.1] | 49.4 [38.5 to 60.3]
  At week 28 | 75.6 [66.3 to 84.9] | 50.6 [39.7 to 61.5]
  At week 32 | 72 [62.2 to 81.7] | 46.9 [36 to 57.8]
  At week 36 | 68.3 [58.2 to 78.4] | 43.2 [32.4 to 54]
  At week 40 | 68.3 [58.2 to 78.4] | 38.3 [27.7 to 48.9]
  At week 44 | 63.4 [53 to 73.8] | 37 [26.5 to 47.6]
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; at week 16; Test type: Superiority; p = 0.568, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.59 to 2.65]
Statistical Analysis 2: Comparison: Baricitinib vs Placebo; at week 20; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.92, 95% CI 2-sided [1.40 to 6.09]
Statistical Analysis 3: Comparison: Baricitinib vs Placebo; at week 24; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.38, 95% CI 2-sided [2.10 to 9.15]
Statistical Analysis 4: Comparison: Baricitinib vs Placebo; at week 28; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 3.09, 95% CI 2-sided [1.51 to 6.32]
Statistical Analysis 5: Comparison: Baricitinib vs Placebo; at week 32; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.47 to 6.11]
Statistical Analysis 6: Comparison: Baricitinib vs Placebo; at week 36; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.44 to 5.60]
Statistical Analysis 7: Comparison: Baricitinib vs Placebo; at week 40; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.49, 95% CI 2-sided [1.74 to 6.97]
Statistical Analysis 8: Comparison: Baricitinib vs Placebo; at week 44; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.87, 95% CI 2-sided [1.46 to 5.66]

4. Secondary Outcome: Percentage of Participants Achieving PedACR70 Responder Index
Description: The PedACR70 response is defined as at least 70% improvement from baseline in 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by > 30%. The 6 core response variables included in the PedACR criteria are: Number of active joints (defined as a joint that is swollen or in the absence of swelling has loss of passive motion accompanied by either pain on motion or joint tenderness) in 73 joints, Number of joints with limited range of motion in 69 joints, Physician's Global Assessment of Disease Activity (21-circle VAS), Parent's Global Assessment of Patient's Overall Well-being, Physical function as assessed by the CHAQ and Acute-phase reactant (hsCRP and ESR). When PedACR response is analyzed as secondary endpoint, ESR measure is only used as acute-phase reactant in the core criteria.
Time Frame: Week 16, 20, 24, 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for PedACR70 at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 16 | 54.9 [44.1 to 65.6] | 54.3 [43.5 to 65.2]
  At week 20 | 68.3 [58.2 to 78.4] | 45.7 [34.8 to 56.5]
  At week 24 | 59.8 [49.1 to 70.4] | 37.0 [26.5 to 47.6]
  At week 28 | 67.1 [56.9 to 77.2] | 39.5 [28.9 to 50.2]
  At week 32 | 57.3 [46.6 to 68] | 35.8 [25.4 to 46.2]
  At week 36 | 61 [50.4 to 71.5] | 35.8 [25.4 to 46.2]
  At week 40 | 57.3 [46.6 to 68] | 30.9 [20.8 to 40.9]
  At week 44 | 53.7 [42.9 to 64.5] | 35.8 [25.4 to 46.2]
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; at week 16; Test type: Superiority; p = 0.972, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.52 to 1.87]
Statistical Analysis 2: Comparison: Baricitinib vs Placebo; at week 20; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.27 to 4.81]
Statistical Analysis 3: Comparison: Baricitinib vs Placebo; at week 24; Test type: Superiority; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.33 to 4.97]
Statistical Analysis 4: Comparison: Baricitinib vs Placebo; at week 28; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.57 to 5.94]
Statistical Analysis 5: Comparison: Baricitinib vs Placebo; at week 32; Test type: Superiority; p = 0.009, Regression, Logistic; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.25 to 4.71]
Statistical Analysis 6: Comparison: Baricitinib vs Placebo; at week 36; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.43 to 5.47]
Statistical Analysis 7: Comparison: Baricitinib vs Placebo; at week 40; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.93, 95% CI 2-sided [1.47 to 5.83]
Statistical Analysis 8: Comparison: Baricitinib vs Placebo; at week 44; Test type: Superiority; p = 0.052, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.99 to 3.74]

5. Secondary Outcome: Percentage of Participants Achieving PedACR90 Responder Index
Description: The PedACR90 response is defined as at least 90% improvement from baseline in 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by > 30%. The 6 core response variables included in the PedACR criteria are: Number of active joints (defined as a joint that is swollen or in the absence of swelling has loss of passive motion accompanied by either pain on motion or joint tenderness) in 73 joints, Number of joints with limited range of motion in 69 joints, Physician's Global Assessment of Disease Activity (21-circle VAS), Parent's Global Assessment of Patient's Overall Well-being, Physical function as assessed by the CHAQ and Acute-phase reactant (hsCRP and ESR). When PedACR response is analyzed as secondary endpoint, ESR measure is only used as acute-phase reactant in the core criteria.
Time Frame: Week 16, 20, 24, 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for PedACR90 at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 16 | 29.3 [19.4 to 39.1] | 23.5 [14.2 to 32.7]
  At week 20 | 42.7 [32 to 53.4] | 24.7 [15.3 to 34.1]
  At week 24 | 37.8 [27.3 to 48.3] | 21 [12.1 to 29.9]
  At week 28 | 42.7 [32 to 53.4] | 25.9 [16.4 to 35.5]
  At week 32 | 43.9 [33.2 to 54.6] | 27.2 [17.5 to 36.8]
  At week 36 | 39 [28.5 to 49.6] | 27.2 [17.5 to 36.8]
  At week 40 | 40.2 [29.6 to 50.9] | 23.5 [14.2 to 32.7]
  At week 44 | 42.7 [32 to 53.4] | 23.5 [14.2 to 32.7]
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; at week 16; Test type: Superiority; p = 0.409, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.66 to 2.75]
Statistical Analysis 2: Comparison: Baricitinib vs Placebo; at week 20; Test type: Superiority; p = 0.030, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.07 to 4.23]
Statistical Analysis 3: Comparison: Baricitinib vs Placebo; at week 24; Test type: Superiority; p = 0.022, Regression, Logistic; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.13 to 4.92]
Statistical Analysis 4: Comparison: Baricitinib vs Placebo; at week 28; Test type: Superiority; p = 0.040, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.03 to 4.08]
Statistical Analysis 5: Comparison: Baricitinib vs Placebo; at week 32; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.07 to 4.24]
Statistical Analysis 6: Comparison: Baricitinib vs Placebo; at week 36; Test type: Superiority; p = 0.132, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.85 to 3.42]
Statistical Analysis 7: Comparison: Baricitinib vs Placebo; at week 40; Test type: Superiority; p = 0.050, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.00 to 4.10]
Statistical Analysis 8: Comparison: Baricitinib vs Placebo; at week 44; Test type: Superiority; p = 0.019, Regression, Logistic; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.15 to 4.71]

6. Secondary Outcome: Percentage of Participants Achieving PedACR100 Responder Index
Description: The PedACR100 response is defined as at least 100% improvement from baseline in 3 of any 6 variables in the core set, with no more than 1 of the remaining variables worsening by > 30%. The 6 core response variables included in the PedACR criteria are: Number of active joints (defined as a joint that is swollen or in the absence of swelling has loss of passive motion accompanied by either pain on motion or joint tenderness) in 73 joints, Number of joints with limited range of motion in 69 joints, Physician's Global Assessment of Disease Activity (21-circle VAS), Parent's Global Assessment of Patient's Overall Well-being, Physical function as assessed by the CHAQ and Acute-phase reactant (hsCRP and ESR). When PedACR response is analyzed as secondary endpoint, ESR measure is only used as acute-phase reactant in the core criteria.
Time Frame: Week 16, 20, 24, 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for PedACR100 at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 16 | 14.6 [7 to 22.3] | 17.3 [9 to 25.5]
  At week 20 | 24.4 [15.1 to 33.7] | 19.8 [11.1 to 28.4]
  At week 24 | 18.3 [9.9 to 26.7] | 16 [8.1 to 24]
  At week 28 | 26.8 [17.2 to 36.4] | 19.8 [11.1 to 28.4]
  At week 32 | 28 [18.3 to 37.8] | 21 [12.1 to 29.9]
  At week 36 | 29.3 [19.4 to 39.1] | 21 [12.1 to 29.9]
  At week 40 | 29.3 [19.4 to 39.1] | 17.3 [9 to 25.5]
  At week 44 | 29.3 [19.4 to 39.1] | 16 [8.1 to 24]
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; at week 16; Test type: Superiority; p = 0.620, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.33 to 1.92]
Statistical Analysis 2: Comparison: Baricitinib vs Placebo; at week 20; Test type: Superiority; p = 0.492, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.61 to 2.78]
Statistical Analysis 3: Comparison: Baricitinib vs Placebo; at week 24; Test type: Superiority; p = 0.715, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.50 to 2.75]
Statistical Analysis 4: Comparison: Baricitinib vs Placebo; at week 28; Test type: Superiority; p = 0.384, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.66 to 2.99]
Statistical Analysis 5: Comparison: Baricitinib vs Placebo; at week 32; Test type: Superiority; p = 0.311, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.70 to 3.10]
Statistical Analysis 6: Comparison: Baricitinib vs Placebo; at week 36; Test type: Superiority; p = 0.231, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.75 to 3.34]
Statistical Analysis 7: Comparison: Baricitinib vs Placebo; at week 40; Test type: Superiority; p = 0.129, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.84 to 3.95]
Statistical Analysis 8: Comparison: Baricitinib vs Placebo; at week 44; Test type: Superiority; p = 0.043, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.02 to 4.84]

7. Secondary Outcome: Percentage of Participants With Inactive Disease
Description: Inactive disease is defined as the presence of all of the following:
  1. No joints with active arthritis based on Juvenile Arthritis Disease Activity Score (JADAS) - 27 score,
  2. No fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to JIA as assessed by the investigator,
  3. No active uveitis as assessed by the investigator,
  4. Normal ESR or hsCRP (i.e., within normal limits in the local laboratory or, if elevated, not attributable to JIA),
  5. Physician's Global Assessment of Disease Activity indicating no active disease (Score ranges are 0 to 100 and best possible score on scale is 0) and
  6. Duration of morning stiffness ≤15 minutes.
Time Frame: Week 16, 20, 24, 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for inactive disease at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 16 | 12.2 [5.1 to 19.3] | 11.1 [4.3 to 18.0]
  At week 20 | 13.4 [6.0 to 20.8] | 17.3 [9 to 25.5]
  At week 24 | 17.1 [8.9 to 25.2] | 17.3 [9.0 to 25.5]
  At week 28 | 20.7 [12.0 to 29.5] | 13.6 [6.1 to 21.0]
  At week 32 | 22.0 [13.0 to 30.9] | 13.6 [6.1 to 21.0]
  At week 36 | 23.2 [14.0 to 32.3] | 16.0 [8.1 to 24]
  At week 40 | 20.7 [12.0 to 29.5] | 12.3 [5.2 to 19.5]
  At week 44 | 23.2 [14.0 to 32.3] | 13.6 [6.1 to 21.0]
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; at week 16; Test type: Superiority; p = 0.853, Regression, Logistic; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.40 to 2.98]
Statistical Analysis 2: Comparison: Baricitinib vs Placebo; at week 20; Test type: Superiority; p = 0.432, Regression, Logistic; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.29 to 1.71]
Statistical Analysis 3: Comparison: Baricitinib vs Placebo; at week 24; Test type: Superiority; p = 0.960, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.41 to 2.31]
Statistical Analysis 4: Comparison: Baricitinib vs Placebo; at week 28; Test type: Superiority; p = 0.215, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.73 to 4.01]
Statistical Analysis 5: Comparison: Baricitinib vs Placebo; at week 32; Test type: Superiority; p = 0.173, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.77 to 4.22]
Statistical Analysis 6: Comparison: Baricitinib vs Placebo; at week 36; Test type: Superiority; p = 0.367, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.64 to 3.33]
Statistical Analysis 7: Comparison: Baricitinib vs Placebo; at week 40; Test type: Superiority; p = 0.162, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.77 to 4.67]
Statistical Analysis 8: Comparison: Baricitinib vs Placebo; at week 44; Test type: Superiority; p = 0.113, Regression, Logistic; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.85 to 4.50]

8. Secondary Outcome: Percentage of Participants With Minimal Disease Activity
Description: Minimal disease activity is calculated based on the scores from the
  1. Physician's Global Assessment of Disease Activity
  2. Parent's Global Assessment of Well-Being and
  3. the number of swollen joints. If the physician's global assessment of disease activity is ≤3.5 (score range: 0-100), the parent's global rating of patient's overall well-being is ≤2.5 (score range: 0-100), and the swollen joint count is ≤1 (score range: 0-73), then the participant reaches minimal disease activity. if not, minimal disease activity is not reached.
Time Frame: Week 16, 20, 24, 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for minimum disease activity at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 16 | 36.6 [26.2 to 47] | 40.7 [30 to 51.4]
  At week 20 | 46.3 [35.5 to 57.1] | 33.3 [23.1 to 43.6]
  At week 24 | 43.9 [33.2 to 54.6] | 34.6 [24.2 to 44.9]
  At week 28 | 45.1 [34.4 to 55.9] | 33.3 [23.1 to 43.6]
  At week 32 | 43.9 [33.2 to 54.6] | 32.1 [21.9 to 42.3]
  At week 36 | 40.2 [29.6 to 50.9] | 33.3 [23.1 to 43.6]
  At week 40 | 43.9 [33.2 to 54.6] | 32.1 [21.9 to 42.3]
  At week 44 | 43.9 [33.2 to 54.6] | 27.2 [17.5 to 36.8]
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; at week 16; Test type: Superiority; p = 0.511, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.42 to 1.55]
Statistical Analysis 2: Comparison: Baricitinib vs Placebo; at week 20; Test type: Superiority; p = 0.145, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.84 to 3.20]
Statistical Analysis 3: Comparison: Baricitinib vs Placebo; at week 24; Test type: Superiority; p = 0.349, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.70 to 2.72]
Statistical Analysis 4: Comparison: Baricitinib vs Placebo; at week 28; Test type: Superiority; p = 0.167, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.82 to 3.25]
Statistical Analysis 5: Comparison: Baricitinib vs Placebo; at week 32; Test type: Superiority; p = 0.212, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.78 to 3.07]
Statistical Analysis 6: Comparison: Baricitinib vs Placebo; at week 36; Test type: Superiority; p = 0.577, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.62 to 2.39]
Statistical Analysis 7: Comparison: Baricitinib vs Placebo; at week 40; Test type: Superiority; p = 0.225, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.78 to 2.95]
Statistical Analysis 8: Comparison: Baricitinib vs Placebo; at week 44; Test type: Superiority; p = 0.055, Regression, Logistic; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.98 to 3.90]

9. Secondary Outcome: Percentage of Participants in Remission
Description: Remission is defined as inactive disease for at least 24 consecutive weeks. Inactive disease is defined as the presence of all of the following: 1) No joints with active arthritis based on Juvenile Arthritis Disease Activity Score (JADAS)-27 score, 2) No fever, rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to JIA as assessed by the investigator, 3) No active uveitis as assessed by the investigator, 4) Normal ESR or hsCRP (i.e., within normal limits in the local laboratory or, if elevated, not attributable to JIA), 5) Physician's Global Assessment of Disease Activity indicating no active disease (best possible score on scale [0]) and 6) Duration of morning stiffness ≤15 minutes.
Time Frame: Week 28, 32, 36, 40 and 44
Population: DBW Population: All randomized participants from the DBW period who had data for remission at given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 81
Percentage of participants
  At week 28 | 0 [0 to 0] | 0 [0 to 0]
  At week 32 | 0 [0 to 0] | 1.2 [0 to 3.6]
  At week 36 | 1.2 [0 to 3.6] | 4.9 [0.2 to 9.7]
  At week 40 | 2.4 [0 to 5.8] | 3.7 [0 to 7.8]
  At week 44 | 3.7 [0 to 7.7] | 3.7 [0 to 7.8]

10. Secondary Outcome: Change From Baseline in Juvenile Arthritis Disease Activity Score-27 (JADAS-27) Score
Description: The JADAS-27 score is based on 4 components: 1) Physician's global assessment of disease activity on a 0-100 mm VAS, 2) Parent's global assessment of overall well-being on a 0-100 mm VAS, 3) normalized ESR and 4) number of joints (maximum of 27) with active arthritis (cervical spine, elbows, wrists, metacarpophalangeal joints [from first to third], proximal interphalangeal joints, hips, knees, and ankles). The scores for the each of the first 3 components range from 0 -10; the score for the final component ranges from 0-27. The overall JADAS-27 score is sum of the 4 components and it ranges from 0-57. A higher score indicates more disease activity. Least square (LS) mean was calculated using Analysis of covariance (ANCOVA) model which includes treatment, baseline, prior biologic JIA therapy, combined JIA category and predose exposure ESR category value as fixed factors.
Time Frame: Baseline, Week 44
Population: DBW Population: All randomized participants from the DBW period who had data for at least one post-baseline JADAS-27 score at given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 80 | 78
score on a scale | -14.24 (1.006) | -9.91 (1.013)
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; Test type: Superiority; p = 0.001, ANCOVA; LS Mean difference = -4.33, 95% CI 2-sided [-6.95 to -1.70], Standard Error of Mean 1.328

11. Secondary Outcome: Change From Baseline in Arthritis-Related Pain Severity as Measured by the Childhood Health Assessment Questionnaire (CHAQ) Pain Visual Analog Scale (VAS) Item
Description: CHAQ assesses the health status and physical function of children with juvenile arthritis over the past week. The CHAQ consists of a Disability Index and a Discomfort Index. The disability index consisted of 30 items grouped into the following 8 domains: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each item is scored from 0 to 3 (0 = no difficulty; 1 = some difficulty; 2 = much difficulty and 3 = unable to do or not applicable). The scores of 8 domains were averaged to calculate the CHAQ-Disability Index total score. A higher score indicates worse physical function. The discomfort index consisted of Parent's Global Assessment of Well-Being and pain assessment due to illness. The intensity of pain is scored on a VAS scale ranging from 0-100 mm, with zero referring to "no pain" and 100 referring to "very severe pain". A higher score indicates a worse outcome.
Time Frame: Baseline, Week 44
Population: DBW Population: All randomized participants from the DBW period who had data for at least one post-baseline CHAQ Pain VAS Item at given time point. LS mean was calculated using Analysis of covariance (ANCOVA) model which includes treatment, baseline, prior biologic JIA therapy, combined JIA category and predose exposure ESR category value as fixed factors.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 82 | 79
score on a scale | -29.65 (3.276) | -16.68 (3.202)
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; Test type: Superiority; p = 0.003, ANCOVA; LS Mean difference = -12.97, 95% CI 2-sided [-21.39 to -4.55], Standard Error of Mean 4.262

12. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk and legs); each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area * area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). LS mean was calculated using ANCOVA model which includes treatment, baseline, prior biologic JIA therapy, combined JIA category and predose exposure ESR category value as fixed factors.
Time Frame: Baseline, Week 44
Population: DBW Population: All randomized participants from the DBW period who had at least one post-baseline juvenile psoriatic arthritis (JPsA) were included in this population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 4 | 3
score on a scale | -1.14 (0.291) | -0.79 (0.354)
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; Test type: Superiority; p = 0.574, ANCOVA; LS Mean difference = -0.35, 95% CI 2-sided [-2.62 to 1.91], Standard Error of Mean 0.526

13. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Index
Description: The SPARCC enthesitis is an index used to measure the severity of enthesitis (sites at which tendons and ligaments attach to bones). The SPARCC assesses 16 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include Medial epicondyle (left/right [L/R]), Lateral epicondyle (L/R), Supraspinatus insertion into greater tuberosity of humerus (L/R), Greater trochanter (L/R), Quadriceps insertion into superior border of patella (L/R), Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R), Achilles tendon insertion into calcaneum (L/R), and Plantar fascia insertion into calcaneum (L/R). The SPARCC is the sum of all site scores (range 0 to 16). Higher scores indicate more severe enthesitis. LS mean was calculated using ANCOVA model which includes treatment, baseline, prior biologic JIA therapy, combined JIA category and predose exposure ESR category value as fixed factors.
Time Frame: Baseline, Week 44
Population: DBW Population: All randomized participants from the DBW period who had enthesitis-related juvenile idiopathic arthritis (ERA) or JPsA were included in this population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 19 | 22
score on a scale | -1.51 (0.276) | -1.95 (0.241)
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; Test type: Superiority; p = 0.208, ANCOVA; LS Mean difference = 0.45, 95% CI 2-sided [-0.26 to 1.15], Standard Error of Mean 0.348

14. Secondary Outcome: Change From Baseline in Juvenile Spondyloarthritis Disease Activity (JSpADA) Index
Description: The JSpADA index is used to evaluate the disease activity of juvenile spondyloarthritis. The JSpADA index scores will be determined by following 8 components: active joint count, active enthesitis count, pain over the past week, CRP level related to juvenile spondyloarthritis activity, morning stiffness greater than 15 minutes, clinical sacroiliitis, uveitis and back mobility. All items are transformed to values of 0, 0.5, or 1, and the total score ranges from 0 to 8, where higher scores indicate more disease activity. LS mean was calculated using ANCOVA model which includes treatment, baseline, prior biologic JIA therapy, combined JIA category and predose exposure ESR category value as fixed factors.
Time Frame: Baseline, Week 44
Population: DBW Population: All randomized participants from the DBW period who had ERA or JPsA were included in this population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Baricitinib | Placebo
Number analyzed (Participants) | 15 | 18
score on a scale | -2.56 (0.347) | -1.47 (0.296)
Statistical Analysis 1: Comparison: Baricitinib vs Placebo; Test type: Superiority; p = 0.019, ANCOVA; LS Mean difference = -1.08, 95% CI 2-sided [-1.98 to -0.19], Standard Error of Mean 0.438

15. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Baricitinib Concentration at Steady-State (Cmax, ss)
Description: Maximum Plasma Baricitinib Concentration at Steady-State
Time Frame: For Safety/PK period: Day 1, Day 4, Day 14 (pre dose) and Day 14 (post dose). For OLLI period: Day 1, Day 14, Day 28, Day 56 and 84 (pre dose)
Population: Safety/PK and OLLI population: All randomized participants from the Safety/PK and OLLI periods who had data for Cmax, ss at given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Groups:
- 12 to <18 Years 4-mg QD: Participants aged 12 to <18 years were given 4-mg baricitinib once daily.
- 9 to <12 Years 4-mg QD: Participants aged 9 to <12 years were given 4-mg baricitinib once daily.
- 6 to <9 Years 2-mg QD: Participants aged 6 to <9 years were given 2-mg baricitinib once daily.
- 2 to <6 Years 2-mg QD: Participants aged 2 to <6 years were given 2-mg baricitinib once daily.
Arm/Group | 12 to <18 Years 4-mg QD | 9 to <12 Years 4-mg QD | 6 to <9 Years 2-mg QD | 2 to <6 Years 2-mg QD
Number analyzed (Participants) | 172 | 27 | 8 | 6
Nanograms per milliliter (ng/mL) | 57.7 (28) | 79 (33) | 56.8 (22) | 87.4 (38)

16. Secondary Outcome: PK: Area Under the Baricitinib Concentration-Time Curve During a Dosing Interval at Steady-State (AUCτ,ss)
Description: Area under the concentration-time curve of Baricitinib during a dosing interval at steady state.
Time Frame: as for outcome 15
Population: Safety/PK and OLLI population: All randomized participants from the Safety/PK assessment and OLLI period who had data for AUCτ,ss at given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/millilitre (h*ng/mL)
Arm/Group | 12 to <18 Years 4-mg QD | 9 to <12 Years 4-mg QD | 6 to <9 Years 2-mg QD | 2 to <6 Years 2-mg QD
Number analyzed (Participants) | 172 | 29 | 8 | 6
hour*nanogram/millilitre (h*ng/mL) | 386 (45) | 500 (57) | 254 (27) | 410 (57)

17. Secondary Outcome: Change From Baseline in Immunoglobulin Levels
Description: Change from baseline in Serum Immunoglobulin A, Serum Immunoglobulin G and Serum Immunoglobulin M levels at week 12 are presented.
Time Frame: Baseline, Week 12
Population: Safety/PK and OLLI population: All randomized participants from the Safety/PK and OLLI periods who had data for for at least one post-baseline immunoglobulin levels at given time point.
Measure: Mean (Standard Deviation); unit: Milligrams per decilitre (mg/dL)
Arm/Group | Baricitinib
Number analyzed (Participants) | 220
Milligrams per decilitre (mg/dL)
  Serum Immunoglobulin A: number analyzed (Participants) | 185
  Serum Immunoglobulin A | -15.98 (39.501)
  Serum Immunoglobulin G: number analyzed (Participants) | 189
  Serum Immunoglobulin G | -81.46 (209.549)
  Serum Immunoglobulin M: number analyzed (Participants) | 190
  Serum Immunoglobulin M | -9.86 (26.680)

18. Secondary Outcome: Number of Participants With Change of Immunoglobulin G (IgG) Titers
Description: Number of participants with change of IgG titers eligible for tetanus / diphtheria / acellular pertussis (tDaP) vaccine and pneumococcal conjugate are presented. Participants who were immunized with tDaP or pneumococcal conjugate vaccine had their IgG antibody titers to the antigens evaluated preimmunization and at 4 and 12 weeks postimmunization. A primary immune response was assessed in participants who had never received tDaP or pneumococcal conjugate vaccines previously and secondary/booster responses were assessed if the participants had previously received the vaccines. For pneumococcal conjugate vaccine, number of participants with >= 2-fold increase from baseline in >=6 pneumococcal serotypes at week 4 and 12 is presented. For tDaP vaccine, number of participants with >= 4-fold increase from baseline in participants with baseline titer >=0.1 IU/mL at week 4 and 12 is presented.
Time Frame: Pre-Vaccination to 4 and 12 Weeks Post-Vaccination
Population: Safety/PK and OLLI population: All randomized participants from the Safety/PK assessment and OLLI period who had data for IgG titers at given time point.
Measure: Number; unit: participants
Arm/Group | Baricitinib
Number analyzed (Participants) | 7
participants
  Tetanus toxoid containing vaccine at week 4: number analyzed (Participants) | 4
  Tetanus toxoid containing vaccine at week 4 | 2
  Tetanus toxoid containing vaccine at week 12: number analyzed (Participants) | 3
  Tetanus toxoid containing vaccine at week 12 | 2
  Diphtheria toxoid containing vaccine at week 4: number analyzed (Participants) | 4
  Diphtheria toxoid containing vaccine at week 4 | 2
  Diphtheria toxoid containing vaccine at week 12: number analyzed (Participants) | 3
  Diphtheria toxoid containing vaccine at week 12 | 1
  Pertussis toxin containing vaccine at week 4: number analyzed (Participants) | 4
  Pertussis toxin containing vaccine at week 4 | 2
  Pertussis toxin containing vaccine at week 12: number analyzed (Participants) | 3
  Pertussis toxin containing vaccine at week 12 | 2
  pneumococcal conjugate vaccine at week 4: number analyzed (Participants) | 4
  pneumococcal conjugate vaccine at week 4 | 3
  pneumococcal conjugate vaccine at week 12: number analyzed (Participants) | 3
  pneumococcal conjugate vaccine at week 12 | 2

19. Secondary Outcome: Number of Participants With Product Acceptability and Palatability Assessment
Description: The questionnaire for product acceptability and palatability assessed the participants ability to swallow the tablet, experience relating to the taste, smell and ease of administering and taking the suspension. The questionnaire contained following Questions: Question 1) How did you (your child) like the taste of the medicine? Question 2) How did you (your child) like the smell of the medicine? Question 3) How easy was it for you (your child) to take the medicine today? Question 4) How easy was it for you to use the oral syringe to give your child the dose today? and Question 5) How easy was it for you (your child) to swallow the medicine today? Responses: Liked Very Much, Liked, Neither Liked nor Disliked, Disliked, Disliked Very Much, Very Easy, Easy, Neither Easy nor Hard, Difficult (or Hard) and Very Difficult (or Hard). The number of participants with these responses are presented. Data is presented as "Question Number-Response-Time point".
Time Frame: Baseline and week 12
Population: Safety/PK and OLLI population: All randomized participants from the Safety/PK assessment and OLLI period who had data for product acceptability and palatability at given time point.
Measure: Number; unit: participants
Arm/Group | Baricitinib
Number analyzed (Participants) | 220
participants
  Question 1- Liked Very Much: Baseline: number analyzed (Participants) | 13
  Question 1- Liked Very Much: Baseline | 2
  Question 1- Liked Very Much: Week 12: number analyzed (Participants) | 10
  Question 1- Liked Very Much: Week 12 | 6
  Question 1- Liked: Baseline: number analyzed (Participants) | 13
  Question 1- Liked: Baseline | 8
  Question 1- Liked: Week 12: number analyzed (Participants) | 10
  Question 1- Liked: Week 12 | 2
  Question 1- Neither Liked nor Disliked: Baseline: number analyzed (Participants) | 13
  Question 1- Neither Liked nor Disliked: Baseline | 3
  Question 1- Neither Liked nor Disliked: Week 12: number analyzed (Participants) | 10
  Question 1- Neither Liked nor Disliked: Week 12 | 1
  Question 1- Disliked: Baseline: number analyzed (Participants) | 13
  Question 1- Disliked: Baseline | 0
  Question 1- Disliked: Week 12: number analyzed (Participants) | 10
  Question 1- Disliked: Week 12 | 1
  Question 1- Disliked Very Much: Baseline: number analyzed (Participants) | 13
  Question 1- Disliked Very Much: Baseline | 0
  Question 1- Disliked Very Much: Week 12: number analyzed (Participants) | 10
  Question 1- Disliked Very Much: Week 12 | 0
  Question 2- Liked Very Much: Baseline: number analyzed (Participants) | 13
  Question 2- Liked Very Much: Baseline | 3
  Question 2- Liked Very Much: Week 12: number analyzed (Participants) | 10
  Question 2- Liked Very Much: Week 12 | 2
  Question 2- Liked: Baseline: number analyzed (Participants) | 13
  Question 2- Liked: Baseline | 7
  Question 2- Liked: Week 12: number analyzed (Participants) | 10
  Question 2- Liked: Week 12 | 4
  Question 2- Neither Liked nor Disliked: Baseline: number analyzed (Participants) | 13
  Question 2- Neither Liked nor Disliked: Baseline | 3
  Question 2- Neither Liked nor Disliked: Week 12: number analyzed (Participants) | 10
  Question 2- Neither Liked nor Disliked: Week 12 | 2
  Question 2- Disliked: Baseline: number analyzed (Participants) | 13
  Question 2- Disliked: Baseline | 0
  Question 2- Disliked: Week 12: number analyzed (Participants) | 10
  Question 2- Disliked: Week 12 | 1
  Question 2- Disliked Very Much: Baseline: number analyzed (Participants) | 13
  Question 2- Disliked Very Much: Baseline | 0
  Question 2- Disliked Very Much: Week 12: number analyzed (Participants) | 10
  Question 2- Disliked Very Much: Week 12 | 1
  Question 3- Very Easy: Baseline: number analyzed (Participants) | 13
  Question 3- Very Easy: Baseline | 8
  Question 3- Very Easy: Week 12: number analyzed (Participants) | 10
  Question 3- Very Easy: Week 12 | 7
  Question 3- Easy: Baseline: number analyzed (Participants) | 13
  Question 3- Easy: Baseline | 3
  Question 3- Easy: Week 12: number analyzed (Participants) | 10
  Question 3- Easy: Week 12 | 2
  Question 3- Neither Easy nor Hard: Baseline: number analyzed (Participants) | 13
  Question 3- Neither Easy nor Hard: Baseline | 1
  Question 3- Neither Easy nor Hard: Week 12: number analyzed (Participants) | 10
  Question 3- Neither Easy nor Hard: Week 12 | 0
  Question 3- Difficult (or Hard): Baseline: number analyzed (Participants) | 13
  Question 3- Difficult (or Hard): Baseline | 0
  Question 3- Difficult (or Hard): Week 12: number analyzed (Participants) | 10
  Question 3- Difficult (or Hard): Week 12 | 1
  Question 3- Very Difficult (or Hard): Baseline: number analyzed (Participants) | 13
  Question 3- Very Difficult (or Hard): Baseline | 1
  Question 3- Very Difficult (or Hard): Week 12: number analyzed (Participants) | 10
  Question 3- Very Difficult (or Hard): Week 12 | 0
  Question 4- Very Easy: Baseline: number analyzed (Participants) | 11
  Question 4- Very Easy: Baseline | 5
  Question 4- Very Easy: Week 12: number analyzed (Participants) | 10
  Question 4- Very Easy: Week 12 | 8
  Question 4- Easy: Baseline: number analyzed (Participants) | 11
  Question 4- Easy: Baseline | 6
  Question 4- Easy: Week 12: number analyzed (Participants) | 10
  Question 4- Easy: Week 12 | 2
  Question 4- Neither Easy nor Hard: Baseline: number analyzed (Participants) | 11
  Question 4- Neither Easy nor Hard: Baseline | 0
  Question 4- Neither Easy nor Hard: Week 12: number analyzed (Participants) | 10
  Question 4- Neither Easy nor Hard: Week 12 | 0
  Question 4- Difficult (or Hard): Baseline: number analyzed (Participants) | 11
  Question 4- Difficult (or Hard): Baseline | 0
  Question 4- Difficult (or Hard): Week 12: number analyzed (Participants) | 10
  Question 4- Difficult (or Hard): Week 12 | 0
  Question 4- Very Difficult (or Hard): Baseline: number analyzed (Participants) | 11
  Question 4- Very Difficult (or Hard): Baseline | 0
  Question 4- Very Difficult (or Hard): Week 12: number analyzed (Participants) | 10
  Question 4- Very Difficult (or Hard): Week 12 | 0
  Question 5- Very Easy: Baseline: number analyzed (Participants) | 203
  Question 5- Very Easy: Baseline | 146
  Question 5- Very Easy: Week 12: number analyzed (Participants) | 159
  Question 5- Very Easy: Week 12 | 120
  Question 5- Easy: Baseline: number analyzed (Participants) | 203
  Question 5- Easy: Baseline | 39
  Question 5- Easy: Week 12: number analyzed (Participants) | 159
  Question 5- Easy: Week 12 | 34
  Question 5- Neither Easy nor Hard: Baseline: number analyzed (Participants) | 203
  Question 5- Neither Easy nor Hard: Baseline | 14
  Question 5- Neither Easy nor Hard: Week 12: number analyzed (Participants) | 159
  Question 5- Neither Easy nor Hard: Week 12 | 5
  Question 5- Difficult (or Hard): Baseline: number analyzed (Participants) | 203
  Question 5- Difficult (or Hard): Baseline | 3
  Question 5- Difficult (or Hard): Week 12: number analyzed (Participants) | 159
  Question 5- Difficult (or Hard): Week 12 | 0
  Question 5- Very Difficult (or Hard): Baseline: number analyzed (Participants) | 203
  Question 5- Very Difficult (or Hard): Baseline | 1
  Question 5- Very Difficult (or Hard): Week 12: number analyzed (Participants) | 159
  Question 5- Very Difficult (or Hard): Week 12 | 0

ADVERSE EVENTS:
Time Frame: Baseline through Follow-up (Up To 341 Days)
Description: All participants who received at least one dose of study drug.
Groups:
- Baricitinib PK and OLLI: During the PK/safety and OLLI periods, baricitinib was administered once daily (QD) as a 4-mg for adolescent participants (12 to <18 years of age) and children ≥9 years of age; and 2 mg for children <9 years of age. Participants <6 years of age received an oral suspension. Participants ≥6 to <12 years old had the option of receiving an oral suspension. Participants >12 years old were supplied tablets.
- Placebo DBW: Participants received placebo matched to baricitinib during the DBW period.
- Baricitinib DBW: During the DBW period, baricitinib was administered once daily (QD) as a 4-mg for adolescent participants (12 to <18 years of age) and children ≥9 years of age; and 2 mg for children <9 years of age. Participants <6 years of age received an oral suspension. Participants ≥6 to <12 years old had the option of receiving an oral suspension. Participants >12 years old were supplied tablets.
Arm/Group | Baricitinib PK and OLLI | Placebo DBW | Baricitinib DBW
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 6/220 | 3/81 | 4/82
Other Adverse Events (participants affected / at risk) | 48/220 | 10/81 | 26/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib PK and OLLI (N=220) | Placebo DBW (N=81) | Baricitinib DBW (N=82)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baricitinib PK and OLLI (N=220) | Placebo DBW (N=81) | Baricitinib DBW (N=82)
Nasopharyngitis (Infections and infestations) | 19 (20) | 3 (3) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 1 (1) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15) | 3 (4) | 6 (6)
Headache (Nervous system disorders) | 14 (16) | 3 (3) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT03773978/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03773978/SAP_001.pdf